CLINICAL TRIAL: NCT04123899
Title: An Open-Label, Randomized, Two-sequence, Two-period, Fasting Condition, Single Oral Dose, Cross-over Study of Bioequivalence of "Gaster®D Tab20mg (Famotidine) (Changed Manufacturer)" and "Gaster®D Tab 20mg (Famotidine) (Unchanged Manufacturer, Announced Reference Drug)" in Healthy, Adult, Human Subjects
Brief Title: BE Study of Gaster®D Tab 20mg (Manufacturer Changed)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIBE2019-19
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Gastroduodenal Ulcer
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IGAD→GSTD (Experimental): IGAD: "Gaster®D Tab 20mg (Famotidine) (Unchanged Manufacturer, Announced Reference Drug)" GSTD: "Gaster®D Tab20mg (Famotidine) (Changed Manufacturer)"
  Interventions: Drug: IGAD→GSTD
- GSTD→IGAD (Experimental): IGAD: "Gaster®D Tab 20mg (Famotidine) (Unchanged Manufacturer, Announced Reference Drug)" GSTD: "Gaster®D Tab20mg (Famotidine) (Changed Manufacturer)"
  Interventions: Drug: GSTD→IGAD

INTERVENTIONS:
Drug: IGAD→GSTD — Drug: IGAD First Period: Single oral administration of 1 tablet of "Gaster®D Tab 20mg (Famotidine) (Unchanged Manufacturer, Announced Reference Drug)"
  Other: Washout period 7 days
  Drug: GSTD Second Period: Single oral administration of 1 tablet of "Gaster®D Tab20mg (Famotidine) (Changed Manufacturer)"
  Arms: IGAD→GSTD
Drug: GSTD→IGAD — Drug: GSTD First Period: Single oral administration of 1 tablet of "Gaster®D Tab20mg (Famotidine) (Changed Manufacturer)"
  Other: Washout period 7 days
  Drug: IGAD Second Period: Single oral administration of 1 tablet of "Gaster®D Tab 20mg (Famotidine) (Unchanged Manufacturer, Announced Reference Drug)"
  Arms: GSTD→IGAD

SUMMARY:
An Open-Label, Randomized, Two-sequence, Two-period, Fasting Condition, Single Oral Dose, Cross-over Study of Bioequivalence of "Gaster®D Tab20mg (Famotidine) (Changed Manufacturer)" and "Gaster®D Tab 20mg (Famotidine) (Unchanged Manufacturer, Announced Reference Drug)" in Healthy, Adult, Human Subjects.

DETAILED DESCRIPTION:
1. Study design: An open-Label, randomized, two-sequence, two-period, fasting condition, single oral dose, cross-over study
2. Administration method:

   The subject should maintain a minimum of 10 hours of empty stomach before administration, and swallow an oral dose of 1 tablets (Famotidine 20 mg) after moistening mouth with 20 mL of water and dissolving completely with saliva on the tongue without water at around 8 a.m. on the day of the test at room temperature. The subject should not chew the drug or break it, but should swallow in whole with water. The difference in administration time between the test subjects is about one minute apart, considering the collection time.
3. Wash out period: 7 days
4. Blood collection time: Before the administration, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 hr after the administration (total 13 times)
5. Analysis: Measurement of the concentration of an unchangeable substance of Famotidine in plasma

ELIGIBILITY:
Inclusion Criteria:

1. A person who aged 19 or older at the time of screening
2. No congenital or chronic diseases or pathological symptoms on screening
3. A person who is judged to be suitable for the study by the investigator based on the clinical laboratory examination
4. BMI of 18 to 30 (BMI calculation: kg/m2)
5. No history of gastrointestinal resection that may affect the absorption of drugs
6. No medical history of mental illness within five years prior to screening
7. A person who has fully understood the contents of the consent form for the study and signed the consent form voluntarily and recorded the date of signature
8. A person who is willing and able to follow all scheduled hospitalization and outpatient visits, medications, clinical laboratory examination and the terms of compliance
9. Female patients who were confirmed to be not pregnant at medical examination

Exclusion Criteria:

1. A person who has taken a drug that significantly induces (e.g., barbital) or inhibits the drug metabolic enzyme within 30 days prior to first administration of the IP
2. A person who uses drugs that can affect the study within 10 days before first administration of the IP
3. A person who is considered unsuitable to participate in the study by the investigator
4. A person who has participated in other clinical trials within 6 months prior to the first administration of the IP
5. A person who has had whole blood transfusion within 2 months or the apheresis within 2 weeks before first administration of IP
6. A person who is hypersensitive to venipuncture
7. A person with a history of regular alcohol intake within six months prior to screening:

   * Women: More than 14 glasses/week
   * Men: More than 21 glasses/week (1 shot: 50 ml of soju, 30 ml of spirits, 250 ml of beer)
8. Blood AST (GOT) or ALT (GPT) levels exceed the upper reference range limit by 2 times or γ-GTP levels exceed the upper reference range limit by 1.5 times
9. Hypersensitive to any of the IP components
10. Patient with hereditary disease Phenylketonuria who need to regulate their intake of phenylalanine
11. Lactating women
12. A person who does not agree to exclude the possibility of pregnancy using the contraception from the date of the first administration of the IP until the 7th day after the last administration.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-10-11 (Estimated); Primary Completion 2019-11-21 (Estimated); Study Completion 2020-01-03 (Estimated)

PRIMARY OUTCOMES:
AUClast | Before administration ~ 24hr
  Area Under the plasma Concentration versus time curve(AUClast) of Famotidine
Cmax | Before administration ~ 24hr
  Peak Plasma Concentration(Cmax) of Famotidine